CLINICAL TRIAL: NCT03038789
Title: XIGDUO Extended Release (XR) (DAPAGLIFLOZIN/METFORMIN XR FDC) Regulatory Postmarketing Surveillance To Observe Safety and Effectiveness Of XigduoXR (Registered) In Korean Patients
Brief Title: XIGDUO Extended Release (XR) Post Marketing Surveillance
Acronym: XigduoPMS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1691R00001
Record Dates: First submitted 2016-12-27; First posted 2017-02-01 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Adult Patients With Type 2 Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a local, prospective, non-interventional, regulatory postmarketing surveillance study. Adult patients with type 2 diabetes mellitus who are initiating Xigduo XR as indicated by the Ministry of Food and Drug Safety (MFDS) will be included.

DETAILED DESCRIPTION:
* Primary objective: Descriptive analysis of the proportion (%) of adverse events (AEs), serious adverse events (SAEs), unexpected adverse events∙adverse drug reactions and AEs of special interest (AESI) in patients who are treated with Xigduo XR for type 2 diabetes mellitus by physicians in the normal clinical practice setting over a period of 12 or 24 weeks.
* Secondary objective: To follow the changes of values of hemoglobin A1c (HbA1c), fasting plasma glucose (FPG), 2-hr post-prandial glucose (PPG-2hr), blood pressure, abdominal circumference and body weight and self-reported data in this cohort of patients from baseline to completion of the study.

To evaluate the safety and tolerability of Xigduo XR in patients with type 2 diabetes mellitus based on conducted laboratory test (Laboratory tests are not mandatory because of the non-interventional nature of this study)

ELIGIBILITY:
Inclusion Criteria:

-Patients will be enrolled by a continuous registration method. Investigators should enroll adult patients who are diagnosed with T2DM and who initiate treatment with Xigduo XR for the first time. Patients (or a legally acceptable representative) who has been informed of all pertinent aspects of the study will sign the Informed Consent Form for use of data. Discontinuation of treatment will be determined by a patient's willingness to continue treatment and the investigator's discretion. The reason for discontinued treatment will be documented.

1. Patients aged 18 years and older
2. Patients with T2DM eligible for treatment with Xigduo XR at first according to the indication as indicated in the locally approved prescribing information
3. Patients with evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

Exclusion Criteria:

1. Hypersensitivity to the active substances or to any of the excipients
2. Patients with renal impairment (e.g., serum creatinine levels ≥ 1.5 mg/dL for men, ≥ 1.4 mg/dL for women, or creatinine clearance < 60 milliliter(mL)/min or estimated glomerular filtration rate (eGFR)< 60mL/min/1.73 m2) which may also result from conditions such as cardiovascular collapse (shock), acute myocardial infarction, and septicemia.
3. Patients with type 1 diabetes mellitus, lactic acidosis, or acute or chronic metabolic acidosis including diabetic ketoacidosis with or without a coma
4. Diabetic precoma
5. Congestive heart failure that medicinal treatment is required
6. Patients with radiologic studies involving the use of intravascular iodinated contrast materials (for example, intravenous urogram, intravenous cholangiography, angiography, and computed tomography (CT) scans with intravascular contrast materials)
7. Patients with severe infection or severe traumatism
8. In terms of Surgical procedures (except minor procedures not associated with restricted intake of food and fluids)
9. Patients with nutrition poor condition, starvation condition, pituitary insufficiency, capsular insufficiency
10. Patients with impaired hepatic function (Since impaired hepatic function has been associated with some cases of lactic acidosis, this drug should generally be avoided in patients with clinical or laboratory evidence of hepatic disease.), respiratory failure, acute myocardial infarction, acute or chronic disease causing histotoxic hypoxia like shock, an alcoholic, gastroenteric trouble (anhydremia, diarrhea, vomiting and etc.)
11. Pregnant women, women with potential of pregnancy, lactating women
12. Patients with hereditary problems such as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients who are diagnosed with type 2 diabetes mellitus (T2DM) eligible for the treatment with Xigduo XR according to prescription information approved by MFDS and as decided by the investigator
Sampling Method: Non-Probability Sample
Enrollment: 623 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Descriptive analysis of the percentage (%) of adverse events (AEs), serious adverse events (SAEs), unexpected adverse events∙adverse drug reactions and AEs of special interest (AESI) | 12 or 24 weeks
  * Percentage (%) of AEs, SAEs and AESI in patients who are treated with Xigduo XR
  * Nature, incidence and severity of AE in patients who are treated with Xigduo XR
  * Nature, incidence and severity of unexpected adverse drug reactions in patients who are treated with Xigduo XR

SECONDARY OUTCOMES:
Hemoglobin A1c (HbA1c) | 12 or 24 weeks
  Change in HbA1c in % during the observation period to evaluate effectivenss
Fasting plasma glucose (FPG) | 12 or 24 weeks
  Change in FPG in mg/dL during the observation period to evaluate effectivenss
2-hr post-prandial glucose (PPG-2hr) | 12 or 24 weeks
  Change of PPG-2hr in mg/dL during the observation period to evaluate effectivenss
Blood pressure | 12 or 24 weeks
  Change in blood pressure in mmHg during the observation period to evaluate effectivenss
Abdominal circumference | 12 or 24 weeks
  Change in abdominal circumference in cm during the observation period to evaluate effectiveness
Body weight | 12 or 24 weeks
  Change in body weight in Kg during the observation period to evaluate effectiveness
Overall investigator's assessment on the outcome of the treatment | 12 or 24 weeks
  Overall investigator's assessment on the outcome of the treatment: "Improved", "Unchanged", "Worsened", "Assessment impossible"
Number of Participants With Abnormal Laboratory Values | 12 or 24 weeks
  Laboratory measures (chemistry/hematology/ urinalysis) during the observation period to evaluate the safety and tolerability of Xigduo XR based on conducted laboratory test (Laboratory tests are not mandatory because of the non-interventional nature of this study).
  * Chemistry: AST, ALT, BUN, Cr, Na+, K+, Total cholesterol, TG
  * Hematology: Hb, Hct
  * Urinalylsis: Proteinurea

CONTACTS AND LOCATIONS:
Overall Officials: JiSeong Yoon, PhD, Principal Investigator — YoungNam University Hospital
Locations (8):
- South Korea (8):
  - Research Site, Busan
  - Research Site, ChungCheong
  - Research Site, Daegu
  - Research Site, Daejeon
  - Research Site, Gyeonggi-do
  - Research Site, Seoul
  - Research Site, Suncheon
  - Research Site, Wŏnju

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: D1691R00001 CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1691R00001&attachmentIdentifier=2678caf3-b8c2-455f-905c-e38a498d516d&fileName=D1691R00001_CSR_synopsis.pdf&versionIdentifier=